CLINICAL TRIAL: NCT00616551
Title: Open Label, Randomized Study Comparing the Biological Efficacy & Safety of a New Prolonged Release Formulation of Octreotide Acetate, C2L-OCT-01 PR, 30 mg Administered Every 42 Days for 84 Days With Sandostatin LAR 30 mg Administered Every 28 Days for 84 Days to Acromegalic Patients
Brief Title: Efficacy and Safety of C2L-OCT-01 PR in Acromegalic Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ambrilia Biopharma, Inc. (Industry)
Responsible Party: Bonabes de Rouge, M.D./Senior Executive Vice-President & Chief Scientist Officer, Ambrilia Biopharma, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C2L-OCT-01 PR-301
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Last update posted 2008-10-08 (Estimated); Status verified 2008-10

CONDITIONS: Acromegaly
Keywords: Acromegaly
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: C2L-OCT-01 PR, 30 mg
- B (Active Comparator)
  Interventions: Drug: Octreotide acetate prolonged release, 30 mg

INTERVENTIONS:
Drug: C2L-OCT-01 PR, 30 mg — Administered by deep IM injection (gluteus) on days 1 and 42
  Arms: A
Drug: Octreotide acetate prolonged release, 30 mg — Administered by deep IM (gluteus) on Days 1, 28 and 56
  Other Names: Sandostatin LAR, 30 mg
  Arms: B

SUMMARY:
The purpose of this study is to assess the biological safety and efficacy of using the drug, C2L-OCT-01 PR, 30 mg to treat acromegalic patients.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be diagnosed with active acromegaly.
* If subject is treated with a long acting somatostatin analogue, the treatment must have been unchanged for a period of at least 12 weeks prior to entry.
* If subject is treated with a 30 mg dose of a depot formulation of a somatostatin analogue, the IGF-1 levels must be normal at entry.
* If subject is treated with a 20 mg dose of a depot formulation of a somatostatin analogue, any value of IGF-1 is acceptable.
* If the subject is receiving an immediate release formulation of a somatostatin analogue or a dopamine agonist, the IGF-1 values must be above 10% of the reference range based on gender and age.
* If the subject is receiving a dopamine agonist, it must be stopped 14 days prior to receiving the study medication.
* The subject should be able to understand the instructions, provide a written consent and abide by the study restrictions.

Exclusion Criteria:

* Women of childbearing potential who are not taking adequate contraception or who are pregnant or lactating.
* Subjects previously treated with a growth hormone receptor antagonist (Pegvisomant) within 12 weeks of study entry.
* Subjects who have undergone pituitary surgery within 6 months or radiotherapy within 2 years prior to admission into the study
* Subjects who present some form of intolerance or allergy to the test article or one of its non-active ingredients
* Subject who have any other condition that alters the growth hormone or IGF-1 levels.
* Subjects with signs or symptoms related to a tumor compression of the optical chiasm.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2007-04; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Compare the mean serum concentrations of insulin-like growth factor-1 (IGF-1) and growth hormone (GH) in patients treated with C2L-OCT-01 PR, 30 mg or Sandostatin LAR 30 mg | Days 1, 28, 42, 56 and 84

SECONDARY OUTCOMES:
Compare plasma concentrations, efficacy and safety profile of C2L-OCT-01 PR | 84 days

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Naudin, M.D., Study Director — Ambrilia Biopharma, Inc.
Locations (6):
- Republican Centre for Medical Rehabilitation and Water-therapy, Minsk, Belarus
- Semmelweis Egyetem Általános Orvostudományi, Budapest, Hungary
- Institute of Endocrinology "C. I. Parhon" Bucharest, Bucharest, Romania
- Institute of Endocrinology, University Clinical Center, Belgrade, Serbia
- Fakultná Nemocnica s Poliklinkou Bratislava, Bratislava, Slovakia
- V.P. Komisarenko Institute of Endocrinology and Metabolism, AMS Ukraine, Kiev, Ukraine